CLINICAL TRIAL: NCT06152536
Title: Effect of a Vegetarian Meal on the Pathophysiology of Insulin Response: a Randomized Controlled Crossover Study in Patients With Type 2 Diabetes and Obesity
Brief Title: Effect of a Vegetarian Meal on the Physiology of Insulin Response in Patients With Type 2 Diabetes Mellitus and Obesity
Acronym: VEG-EAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Emanuele Bosi, Professor, IRCCS San Raffaele
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 04/INT/2022
Record Dates: First submitted 2023-02-14; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Type2diabetes; Obesity; Diet, Healthy; Nutrition, Healthy
Keywords: nutrition; meal; insulin; glycemia
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Monocentric, controlled and randomized trial in crossover.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meal 2 (Experimental): Meal with a vegetarian protein
  Interventions: Other: Vegetarian Meal
- Meal 1 (Active Comparator): Meal with animal protein
  Interventions: Other: Vegetarian Meal

INTERVENTIONS:
Other: Vegetarian Meal — "meal with vegetarian protein" and "meal with animal protein"

SUMMARY:
The role of diet in determining glucose intolerance and its progression towards T2DM has been extensively investigated. A 2017 meta-analysis showed that a vegetarian diet is inversely associated with the risk of developing diabetes. Vegetarians, with the same baseline risk, are half as likely to develop T2DM than those following an omnivorous diet. Therefore, vegetarian nutrition could have important clinical implications in the dietary management of diabetic patients.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the effect of two different isocaloric meals, one vegetarian compared to a conventional Mediterranean-type one (vegetable protein source in the first case and animal in the second case), eaten at lunch, 1÷3 weeks apart, on the pathophysiology of glucose and insulin response. The two meals were elaborated in such a way as to have a superimposable composition.

Study population: 20 patients diagnosed with T2DM and BMI ≥ 30, belonging to the Diabetes and Clinical Nutrition clinic of the IRCCS San Raffaele Hospital.

Study design: single-center, interventional, controlled, randomized crossover.

Procedures: the patients enrolled in the study, for each of the two meals, underwent serial blood tests, before eating lunch (T0) and every 30 minutes, up to 3 hours after the end of the meal itself (T2÷T6).

Collected variables: blood sugar, insulin, c-peptide, HbA1c, total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides, height, weight, waist circumference and blood pressure, visual analogue scale (0-10) for sense of hunger and satiety , meal satisfaction index (0-10).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Diagnosis of T2DM
* In treatment with diet alone or single oral drug metformin
* BMI ≥ 30
* HbA1c between 6.0 and 9.0% (42-75 mmol/mol)
* Signature of the informed consent

Exclusion Criteria:

* History of acute/chronic pancreatitis
* Pancreatic cancer
* Pancreatic surgery
* Renal failure (any stage)
* Liver cirrhosis
* Thyroid disorders (hypothyroidism, hyperthyroidism)
* Patients with weight loss in the last 3 months equal to or greater than 5% of body weight
* Patients on therapy other than metformin monotherapy (insulin, glucagon-like peptide agonists, sulphonylureas, glitazones, dipeptidyl peptidase inhibitors, SGLT2 inhibitors).
* Pregnant or breastfeeding women
* History of severe allergic reaction to any food (anaphylaxis)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-06-09 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Physiopathology of glucose after two different meals | fasting, 30 minutes after meal, 60 minutes after meal, 90 minutes after meal, 120 minutes after meal, 150 minutes after meal, 180 minutes after meal,
  evaluation of glycemic curve after a meal with a vegetarian protein compared to the same evaluation after a meal with an animal protein

SECONDARY OUTCOMES:
Physiopathology of insulin after two different meals | fasting, 30 minutes after meal, 60 minutes after meal, 90 minutes after meal, 120 minutes after meal, 150 minutes after meal, 180 minutes after meal,
  evaluation of insulin curve after a meal with a vegetarian protein compared to the same evaluation after a meal with an animal protein

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fizelova M, Jauhiainen R, Stancakova A, Kuusisto J, Laakso M. Finnish Diabetes Risk Score Is Associated with Impaired Insulin Secretion and Insulin Sensitivity, Drug-Treated Hypertension and Cardiovascular Disease: A Follow-Up Study of the METSIM Cohort. PLoS One. 2016 Nov 16;11(11):e0166584. doi: 10.1371/journal.pone.0166584. eCollection 2016. PMID 27851812